CLINICAL TRIAL: NCT00169611
Title: Comportemental and Neuropsychologic Study of Children With Neurofibromatosis Type 1 Treated by Methylphenidate. A Double-blind Randomised Study Methylphenidate Versus Placebo
Brief Title: NF1-Attention: Study of Children With Neurofibromatosis Type 1 Treated by Methylphenidate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Dr Laurence LION-FRANCOIS, Service de Neuropédiatrie - Hôpital Femme Mère Enfant -
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2003.310
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis type 1; Attention deficit with hyperactivity disorder school difficulties; methylphenidate
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
Neurofibromatosis type 1 (NF1) is an autosomal dominant disorder with an estimated prevalence of 1/2190 to 1/6711. Attention deficit hyperactivity disorder (ADHD) has been reported to be common in NF1. We, the researchers at Hospices Civils de Lyon, designed a randomized, double blind, placebo controlled, crossover trial with a total follow-up duration of 9 weeks to evaluate the effect of methylphenidate (MPH) on the improvement on the simplified parents Conners' Rating Scale. In a parallel exploratory study we will compare the nature of attention deficit disorders in NF1 children to 30 ADHD NF1-free controls. Children aged 7 to 12 years are eligible when their intelligence quotient (IQ) is between 80 and 120. Fifty subjects (25 for each period) were required for testing the primary study hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years
* IQ between 80-120.
* Gender: male or female
* Children with neurofibromatosis type 1 (according to the National Institutes of Health [NIH] 1988).
* Patients with school difficulties pointed out by parents or teachers
* Patients with attention difficulties as defined by anamnesis

Exclusion Criteria:

* IQ > 120 or IQ < 80
* Child depression
* Unwillingness to participate
* Patients with cerebral complication of neurofibromatosis type 1 (chiasma glioma, moya-moya) as detected by cerebral magnetic resonance imaging (MRI).
* Participation in another study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2004-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Effect of methylphenidate compared to placebo on ADHD. Time of measurements are realised on day 0, day 28, day 63 + 2 days.

SECONDARY OUTCOMES:
To evaluate the efficacy of methylphenidate compared to placebo on specific neuropsychologic, depression and anxiety scales
To compare the nature of attention deficit disorders in NF1 children with those with primary ADHD, depression, and anxiety using the State Trait Anxiety Inventory for Children (STAI-C) and the Children's Depression Inventory (CDI).
Time of measurements are realised on day 0, day 28, day 63 + 2 days.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LION-FRANCOIS, MD, Principal Investigator — Service de Neuropédiatrie - Hôpital Femme Mère Enfant - Hospices Civils de Lyon - 59 bd Pinel - 69677 BRON - France; Isabelle KEMLIN, Principal Investigator — Service de Neuropédiatrie - Hôpital Armand Trousseau - PARIS - France
Locations (1):
- Laurence LION-FRANCOIS, Lyon, France

REFERENCES:
- [Derived] Lion-Francois L, Gueyffier F, Mercier C, Gerard D, Herbillon V, Kemlin I, Rodriguez D, Ginhoux T, Peyric E, Coutinho V, Breant V, des Portes V, Pinson S, Combemale P, Kassai B; Reseau NF1 Rhone Alpes Auvergne-France. The effect of methylphenidate on neurofibromatosis type 1: a randomised, double-blind, placebo-controlled, crossover trial. Orphanet J Rare Dis. 2014 Sep 10;9:142. doi: 10.1186/s13023-014-0142-4. PMID 25205361
- See also: Related Info — http://www.orphanet.org